CLINICAL TRIAL: NCT06531304
Title: Patient-therapist INTERaction During RObotic GAIT Rehabilitation After Spinal Cord Injury: Clinical, Instrumental and Hyperscanning Study.
Brief Title: Patient-therapist INTERaction During RObotic GAIT Rehabilitation After Spinal Cord Injury
Acronym: INTERROGAIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Federica Tamburella, Associate Professor, PhT, PhD, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR-2019-12369207
Record Dates: First submitted 2024-07-25; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injuries
Keywords: Physical Therapist-Patient interaction; incomplete SCI; RAGT
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical/Functional evaluation of patients will be performed by expert physiotherapists blinded to group allocation.
  Data analysis (EEG, EMG, Kinematic, Kientic) will be performed by neuroscientists blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXP GROUP (Experimental): Patients will receive visual FB information about the Lokomat joint torque on the screen in front of him/her in order to adapt on-line hips and knees performances. In the EXP group, the Physical Therapist will receives also visual FB information and will guide the patient along the sessions with continuos verbal instructions, thus optimizing the PhT-Pt interaction with an high level of interaction. Patient will be asked to modify his/her hips or knees performances according to both the FB visualized on the screen and the information provided by the PhT.
  Interventions: Device: Lokomat Robot Assisted Gait Training
- CTRL GROUP (Active Comparator): Patients will receive visual FB information about the Lokomat joint torque on the screen in front of him/her in order to adapt on-line hips and knees performances, but the level on interaction between Patient and Physical Therapist will be reduced to its minimum because of no verbal instruction provided by the Physical Therapist to the patient. Consequently, patient will be asked to modify his/her hips or knees performances according only to the FB visualized on the screen, without no technical exchange with the Physical Therapist.
  Interventions: Device: Lokomat Robot Assisted Gait Training

INTERVENTIONS:
Device: Lokomat Robot Assisted Gait Training — Patients will underwent 12 RAGT training sessions (3 times/week for 4 consecutive weeks, 45 min each including the time for wearing the harness and the exoskeleton) with the Lokomat device as add-on to conventional regimen (5 times/week, 80 min each). The Lokomat is a technologically advanced robot-assisted gait training device. Patients are supported in a harness above a treadmill while the robotic device assists the movements of their legs to provide physiological gait. As treatment progresses, weight bearing is increased and assistance from the robotic legs is reduced, requiring the patient to gradually assume greater responsibility for movements needed during walking.

SUMMARY:
INTERROGAIT will disentangle the role of Physical Therapist - Patient (Pht-Pt) interaction in robotic assisted gait rehabilitation in spinal cord injury patients. The study is structured as a single blind randomized controlled trial with two arms, in which effects of different Pht-Pt interaction levels will be assessed on the ongoing robotic treatment with the Lokomat device. The main hypothesis is that when Pht-Pt interaction is maximized (experimental group), this will allow to better rehabilitation outcome with respect to a minimun level of Pht-Pt interaction (control group).

DETAILED DESCRIPTION:
Gait recovery is a main goal in the rehabilitation of individuals with in incomplete SCI (i-SCI). Modern approaches favor task specific repetitive rehabilitation, with high intensity and early multisensorial stimulation such as the robot assisted gait training (RAGT). The growing interest in robotic therapy has attracted attention to human-robot interactions in the rehabilitation framework, and a consensus is forming on the importance of top-down approaches in rehabilitation, particularly when dealing with robotic devices. The critical aspects of top-down approaches are multifarious and include motivation, active participation, learning skills and error-driven-learning, evidencing the key aspects of feedback (FB) information to guide and improve HRI interactions. These evidences highlight the crucial function of active patient (Pt) involvement and the importance of information that is provided by the physiotherapist (PhT) to the Pt for supporting recovery. Further, Pts who feel engaged in the treatment and receive FB are more adherent to rehabilitation and the Pht can provide reinforcement, giving positive attention, praise, and encouragement for the Pt's effort. PhT-Pt interaction is a key aspect for success in rehabilitation: physical, verbal, and technical exchanges between the PhT and Pt highly influence the outcome. In robotic gait rehabilitation Pht-Pt interaction depends on various aspects which include the amount and quality of information exchanged between Pt and robot and Pht and robot, in a threefold relationship.

Recent data on human-to-human interactions and neural correlates of interpersonally coordinated motor behavior have indicated that cooperative motor behavior engages specific cortical and subcortical areas of the motor system compared with execution of the task alone, promoting the learning of motor strategies to support recovery. Recently, a new conceptual and methodological framework has been proposed to investigate the neural basis of human social interaction: the two-person neuroscience. It focuses on studying the dual exchange rather than only on the individual behavior, by using simultaneous neurophysiological recordings from two or more subjects, commonly referred to as hyperscanning or dual scanning. An approach that can provide a viable way to untangle the social interaction from two-persons data is multiple-brain connectivity (also referred to, in some studies, as hyperconnectivity). Thereby temporal correlations between signals derived from the brain regions of different subjects during their interaction are studied to understand how the brain activity of each subject is correlated to the activity in the brain of the other subject. Inter-subject connectivity was described by fMRI, MEG and EEG studies, the latter allowing for an ecological setting. Furthermore, the use of indices derived from graph theory allows to characterize the multiple brain system by means of its properties. The literature is vast on the effects of RAGT on i-SCI gait performances, particularly on speed parameters. However the impact of Pht-Pt interaction on gait outcome has never been investigated in this context at the time of this proposal. The combination of EEG hyperscanning and multiple-brain connectivity could be a powerful tool to objectively measure the Pht-Pt interaction and put it in relation with the rehabilitation outcomes. INTERROGAIT will explore such context by modulating Pht-Pt interaction during gait rehabilitation with the Lokomat device in iSCI patients.

The main hypothesis is that RAGT performed using the FB provided the Lokomat device with an high level of Pht-Pt interaction can lead to a better functional outcome for Pts, in comparison to a minimum interaction. Moreover, we will provide quantitative assessment of Pht-Pt interaction (EEG hyperscanning study) and seek for correlations between neurophysiological descriptors and clinical outcome, supporting our main hypothesis.

The main aim of this study is to test the effects of maximum and minimum PhT-Pt interaction in RAGT on clinical and functional performences in iSCI subjects, through a single blind longitudinal randomized controlled clinical trial.

Furthermore, the study will be aimed to identify neurophysiological indices derived from hyperscanning EEG data monitoring the establishment and development of Pht-Pt interaction during RAGT and to investigate the correlation between the establishment of a successful Pht-Pt interaction as assessed via neurophysiological indices and psychological variables and the rehabilitation outcome. Aspects related to acceptability and usability of the approaches will be evaluated. In detail for the Pt mood, motivation and satisfaction will be evaluated before (mood, motivation) and after (satisfaction) RAGT sessions by means of Visual Analogue Scales; workload will be evaluated at the end of the training sessions by means of the Nasa-Task Load Index. For both Pht and Pt the empathy and the ability to recognize or express emotion will be assesses before and after the training according to Emotional Response Scale, Impression Scale, Interpersonal Reactivity Index,Empathy Quotient, Assertion Inventory, Responsibility Attitude Scale.

ELIGIBILITY:
Inclusion Criteria:

* incomplete SCI lesion (ISNCSCI AIS level C or D);
* subacute or chronic iSCI;
* traumatic and non-traumatic aetiology;
* SCI at or above T12 level;
* absence of severe cognitive impairment such as to interfere with the protocol.

Exclusion Criteria:

* lack of the clinical requirements for using Lokomat;
* anything preventing EEG recording.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in 10 Meters Walking Test (10MWT) | Within 24 h before starting RAGT intervention (Pre) and within 24 hours from the twelfth Lokomat session (Post)
  Time test for gait speed assessment on short distance. The patients are instructed to walk a 10 meters distance, and the gait speed is calculated.
Changes in Min Walking test (6MWT) | Within 24 h before starting RAGT intervention (Pre) and within 24 hours from the twelfth Lokomat session (Post)
  Time test for gait speed assessment on long distance. The distance covered over a time of 6 minutes is recorded, and the gait speed is calculated

SECONDARY OUTCOMES:
Changes in Walking Index for Spinal Cord Injury II (WISCI-II) | Within 24 h before starting RAGT intervention (Pre) and within 24 hours from the twelfth Lokomat session (Post)
  WISCI-II assess the amount of physical assistance needed, as well as devices or orthosis required, for walking following iSCI. Scores range from 0 (inability to walk) and 20 (patient can walk with no assistance, no aids, no orthoses)
Changes in Lower-extremity motor scores (LEMS) of American Spinal Cord Injury Association | Within 24 h before starting RAGT intervention (Pre) and within 24 hours from the twelfth Lokomat session (Post)
  The LEMS evaluates motor function on a scale that ranges from 0 (no motor function) to 5 (full motor function) for 5 lower extremity muscle groups with a 50-point maximum (25 per side). The key muscles of the lower limbs assessed for LEMS are: hip flexor muscles, knee extensor muscles, ankle dorsiflexor muscles, long toe extensors muscles, and ankle plantarflexor muscles.
Changes in Modified Ashworth Scale (MAS) | Within 24 h before starting RAGT intervention (Pre) and within 24 hours from the twelfth Lokomat session (Post)
  The MAS for spasticity assessment is a 6 points numerical scale that graded spasticity from 0 to 4, with 0 being no resistance and 4 being a limb rigid in flexion or extension.
Changes in Independence in activities of daily living per the Spinal Cord Independence Measure III (SCIM-III) | Within 24 h before starting RAGT intervention (Pre) and within 24 hours from the twelfth Lokomat session (Post)
  The SCIM-III is designed for individuals with SCI and assesses performance in activities of daily living and mobility. There are a total of 19 items, which are divided into 3 subscales (self-care, respiration and sphincter management, and mobility). A total score out of 100 is achieved, with the subscales weighted as follows: self-care: scored 0-20; respiration and sphincter management: scored 0-40; and mobility: scored 0-40. Scores are higher in patients that require less assistance or fewer aids to complete basic activities of daily living and life support activities.

OTHER OUTCOMES:
Changes in Patient EEG spectral activity and Pht-Pt inter-brain connectivity | Within 24 h before starting RAGT intervention (Pre) and within 24 hours from the twelfth Lokomat session (Post)
  High density Electroencephalography (hdEEG) signals will be recorded simultaneously (EEG hyperscanning) from Pt and Pht during their interaction. Changes in Pt patterns of cortical oscillatory activity and Pht-Pt inter-brain connectivity, as assessed during neurophysiological assessment before and after the intervention, will be investigated. The analysis will focus on spectral activations of specific brain regions and objective indices characterizing Pht-Pt multiple-brain connectivity patterns within motor related frequency band.
Changes in Kinematic, Kinetic and Electromyography parameters | Within 24 h before starting RAGT intervention (Pre) and within 24 hours from the twelfth Lokomat session (Post)
  Kinematic, Kinetic and surface Electromyography parameters of the lower limbs will be recorded both during gait on a flat surface, to detect at least 5 gait cycles, with the Optitrack system for instrumental gait analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Tamburella, Principal Investigator — I.R.C.C.S. Fondazione Santa Lucia
Locations (1):
- I.R.C.C.S. Fondazione Santa Lucia, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
Clinical and neurophysiological Data (EMG, Kinematic, Kinetic,EEG) will be shared upon reasonable request (anonymized)

REFERENCES:
- [Background] Tamburella F, Moreno JC, Herrera Valenzuela DS, Pisotta I, Iosa M, Cincotti F, Mattia D, Pons JL, Molinari M. Influences of the biofeedback content on robotic post-stroke gait rehabilitation: electromyographic vs joint torque biofeedback. J Neuroeng Rehabil. 2019 Jul 23;16(1):95. doi: 10.1186/s12984-019-0558-0. PMID 31337400
- [Background] Belda-Lois JM, Mena-del Horno S, Bermejo-Bosch I, Moreno JC, Pons JL, Farina D, Iosa M, Molinari M, Tamburella F, Ramos A, Caria A, Solis-Escalante T, Brunner C, Rea M. Rehabilitation of gait after stroke: a review towards a top-down approach. J Neuroeng Rehabil. 2011 Dec 13;8:66. doi: 10.1186/1743-0003-8-66. PMID 22165907
- [Background] Tamburella F, Moreno JC, Iosa M, Pisotta I, Cincotti F, Mattia D, Pons JL, Molinari M. Boosting the traditional physiotherapist approach for stroke spasticity using a sensorized ankle foot orthosis: a pilot study. Top Stroke Rehabil. 2017 Sep;24(6):447-456. doi: 10.1080/10749357.2017.1318340. Epub 2017 May 1. PMID 28460597
- [Background] Koike T, Tanabe HC, Sadato N. Hyperscanning neuroimaging technique to reveal the "two-in-one" system in social interactions. Neurosci Res. 2015 Jan;90:25-32. doi: 10.1016/j.neures.2014.11.006. Epub 2014 Dec 10. PMID 25499683
- [Background] Krill AL, Platek SM. Working together may be better: activation of reward centers during a cooperative maze task. PLoS One. 2012;7(2):e30613. doi: 10.1371/journal.pone.0030613. Epub 2012 Feb 15. PMID 22355319
- [Background] Montague PR, Berns GS. Neural economics and the biological substrates of valuation. Neuron. 2002 Oct 10;36(2):265-84. doi: 10.1016/s0896-6273(02)00974-1. PMID 12383781
- [Background] Babiloni F, Astolfi L. Social neuroscience and hyperscanning techniques: past, present and future. Neurosci Biobehav Rev. 2014 Jul;44:76-93. doi: 10.1016/j.neubiorev.2012.07.006. Epub 2012 Aug 13. PMID 22917915
- [Background] Hari R, Himberg T, Nummenmaa L, Hamalainen M, Parkkonen L. Synchrony of brains and bodies during implicit interpersonal interaction. Trends Cogn Sci. 2013 Mar;17(3):105-6. doi: 10.1016/j.tics.2013.01.003. Epub 2013 Feb 4. PMID 23384658
- [Background] Bilek E et al 2015 PNAS 112: 5207-5212
- [Background] King-Casas B, Tomlin D, Anen C, Camerer CF, Quartz SR, Montague PR. Getting to know you: reputation and trust in a two-person economic exchange. Science. 2005 Apr 1;308(5718):78-83. doi: 10.1126/science.1108062. PMID 15802598
- [Background] Campi C, Parkkonen L, Hari R, Hyvarinen A. Non-linear canonical correlation for joint analysis of MEG signals from two subjects. Front Neurosci. 2013 Jun 14;7:107. doi: 10.3389/fnins.2013.00107. eCollection 2013. PMID 23785311
- [Background] Toppi J, Borghini G, Petti M, He EJ, De Giusti V, He B, Astolfi L, Babiloni F. Investigating Cooperative Behavior in Ecological Settings: An EEG Hyperscanning Study. PLoS One. 2016 Apr 28;11(4):e0154236. doi: 10.1371/journal.pone.0154236. eCollection 2016. PMID 27124558
- [Background] Astolfi L, Toppi J, De Vico Fallani F, Vecchiato G, Cincotti F, Wilke CT, Yuan H, Mattia D, Salinari S, He B, Babiloni F. Imaging the Social Brain by Simultaneous Hyperscanning During Subject Interaction. IEEE Intell Syst. 2011 Oct;26(5):38-45. doi: 10.1109/MIS.2011.61. No abstract available. PMID 22287939
- [Background] Astolfi L, De Vico Fallani F, Cincotti F, Mattia D, Marciani MG, Salinari S, Sweeney J, Miller GA, He B, Babiloni F. Estimation of effective and functional cortical connectivity from neuroelectric and hemodynamic recordings. IEEE Trans Neural Syst Rehabil Eng. 2009 Jun;17(3):224-33. doi: 10.1109/TNSRE.2008.2010472. Epub 2008 Dec 9. PMID 19273037
- [Background] De Vico Fallani F, Nicosia V, Sinatra R, Astolfi L, Cincotti F, Mattia D, Wilke C, Doud A, Latora V, He B, Babiloni F. Defecting or not defecting: how to "read" human behavior during cooperative games by EEG measurements. PLoS One. 2010 Dec 1;5(12):e14187. doi: 10.1371/journal.pone.0014187. PMID 21152069
- [Background] Lindenberger U, Li SC, Gruber W, Muller V. Brains swinging in concert: cortical phase synchronization while playing guitar. BMC Neurosci. 2009 Mar 17;10:22. doi: 10.1186/1471-2202-10-22. PMID 19292892
- [Background] Ciaramidaro A, Toppi J, Casper C, Freitag CM, Siniatchkin M, Astolfi L. Multiple-Brain Connectivity During Third Party Punishment: an EEG Hyperscanning Study. Sci Rep. 2018 May 1;8(1):6822. doi: 10.1038/s41598-018-24416-w. PMID 29717203